CLINICAL TRIAL: NCT01982344
Title: A Study Comparing the Impact of Mini-exchange-room and Usual Care on Physical Activity and Quality of Life in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Institute of Nephrology, Division of Renal, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: mini-exchange-room
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Physical Activity; Quality of Life
Keywords: mini-exchange-room; physical activity; quality of life; peritoneal dialysis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mini-exchange-room (G2) (Experimental): the other group will utilize disposable mini-exchange-room group
  Interventions: Device: mini-exchange-room
- usual care (G1) (No Intervention): The one group perform traditional PD procedure (G1)

INTERVENTIONS:
Device: mini-exchange-room
  Arms: mini-exchange-room (G2)

SUMMARY:
To compare the effect of mini-exchange-room and usual care on physical activity and quality of life in peritoneal dialysis (PD) patients through a randomized controlled study. A total of 80 incident CAPD patients with age of 18~80 years old will be enrolled, who are medically stable and regularly followed up. The one group perform traditional PD procedure (G1), and the other group will utilize disposable mini-exchange-room group (G2). Two groups will be followed for 6 months. Biochemistry data, types of space for bag exchange, physical activity and quality of life will also be collected for all subjects at the 3rd and 6th month. During the study period, peritonitis episode, acute comorbidity and hospitalization will be recorded. The change of physical activity, quality of life and peritonitis rate will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in the Division of Nephrology, Beijing University First Hospital. A total of 80 incident CAPD patients with age of 18~80 years old will be enrolled, who are medically stable and regularly followed up. Informed consent is required for each patient.

Exclusion Criteria:

* Those who have (1) intolerance to the study protocols, (2) severe and unstable conditions within one month, acute or chronic inflammation disease, (3) high probability (assessed by the recruiting physician) of receiving a kidney transplant or transferring to HD or drop-out due to socioeconomic causes within 6 months, (4) cognitive or psychological dysfunction, communication barrier, and (5) bag exchange by unfixed manipulator, are excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
the improvement in physical activity | 6 months
the improvement in quality of life | 6 months

SECONDARY OUTCOMES:
times of bag exchanges outside patients' home | 6 months
peritonitis rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jie Dong, Beijing, Beijing Municipality, China